CLINICAL TRIAL: NCT04375293
Title: Characterisation of the Nasal Microbiome in Patients Suffering From Non-steroidal Anti-inflammatory Drugs-exacerbated Respiratory Disease (N-ERD) - a Pilot Study
Brief Title: Characterisation of the Nasal Microbiome in Patients With N-ERD
Acronym: MicroNERD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Sven Schneider, MD, Principal Investigator, Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: MicroNERD
Record Dates: First submitted 2020-01-24; First posted 2020-05-05 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Aspirin Exacerbated Respiratory Disease; Chronic Rhinitis
Keywords: aerd, microbiome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- AERD (Experimental): Patients suffering from AERD
  Interventions: Other: Microbiome swabs
- Healthy (Sham Comparator): Healthy Controls
  Interventions: Other: Microbiome swabs
- CRSwNP (Active Comparator): Patients suffering from CRS with nasal polyps
  Interventions: Other: Microbiome swabs
- CRSsNP (Active Comparator): Patients suffering from CRS without nasal polyps
  Interventions: Other: Microbiome swabs

INTERVENTIONS:
Other: Microbiome swabs — Swabs for analysis of microbiome

SUMMARY:
Chronic rhinosinusitis (CRS) with (w) and without (s) nasal polyps (NP) in its different shapes is currently affecting up to 16% of the total population of the United States and around 11% of the population in Europe. It may also be associated with a hypersensitivity to non-steroidal anti-inflammatory (NSAID) drugs in a syndrome called NSAID-exacerbated respiratory disease (N-ERD) characterized by highly recurrent polyps and concomitant asthma. The pathophysiological mechanisms especially with regards to the potential role of the microbiome in driving N-ERD are so far not fully understood. Here, the investigators plan to analyse the nasal microbiome in these patients and to compare it to nasal samples from CRSwNP and CRSsNP patients as well as healthy controls (in total 80 subjects). This will provide insights into potential differences in the microbiome as compared to other CRS patients and the impact of the microbiome in driving this disease.

DETAILED DESCRIPTION:
Chronic rhinosinusitis (CRS) with (w) and without (s) nasal polyps (NP) in its different shapes is currently affecting up to 16% of the total population of the United States and around 11% of the population in Europe . However CRS may also be associated with hypersensitivity to aspirin and other non-selective cyclooxygenase inhibitors. This syndrome of combined CRSwNP, asthma and intolerance to inhibitors of the cyclooxygenase-1 enzyme was termed Samter's triad, aspirin-exacerbated respiratory disease (AERD) and recently NSAID-exacerbated respiratory disease (N-ERD). N-ERD is thought to affect around 16% of patients suffering from CRSwNP , around 7% of adult asthmatic patients and 0.3-2.5% of the general population. One characteristic feature of this disease is the presence of nasal polyps that frequently relapse after surgery rendering this disease difficult to manage. Despite its relatively high prevalence, the pathophysiologic mechanisms are yet not fully understood. In this respect, an overproduction of and overresponsiveness to cysteinyl leukotrienes accompanied by and underproduction of and underresponsiveness to prostaglandins was observed in N-ERD patients.This indicates a dysregulation of pro and anti-inflammatory pathways.

Our mucosal body surfaces are colonized by a large variety of microbes organized within complex community structures. Novel sequencing techniques (e.g. 16SrRNA sequencing) have facilitated in-depth analysis of the nasal microbiome in health and disease. Recent studies show amongst other an enrichment in Haemophilus and Streptococcus in the nose of CRS patients, whereas nasal microbiome of healthy patients is rich in Propionibacterium acnes . So far, differences in microbiome were observed in healthy versus CRS patients, but the impact of the microbial environment in N-ERD has not been assessed yet and is thus aim of the study.

The investigators will collect nasal microbiome and nasal secretions from patients suffering from N-ERD and will compare them to the microbiome of CRSwNP, CRSsNP and healthy controls (n=20 per group). Additionally, cytokines in nasal secretions, protein expression at mRNA levels in nasal mucosa, and serum of these patients and clinical parameters (e.g. total nasal polyp score, quality of life questionnaire, olfactory performance) will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Age: 18-90
* Willingness to participate in the study
* No use of nasal or systemic corticosteroids or immunosuppressants 2 weeks prior to their visit
* Patient groups:

  * Control group: absence of any signs of acute or chronic rhinosinusitis
  * CRS:

CRSsNP CRSwNP N-ERD: N-ERD as previously confirmed by clinical history or provocation testing

The presence of CRS will be confirmed by endoscopy (part of routine assessment at the ORL department, no study procedure) according to AAO-HNSF guidelines as follows :

• Twelve weeks or longer of two or more of the following signs and symptoms:

* mucopurulent drainage (anterior, posterior, or both)
* nasal obstruction (congestion)
* facial pain-pressure-fullness, or
* decreased sense of smell

AND inflammation is documented by one or more of the following findings:

* purulent (not clear) mucus or edema in the middle meatus or anterior ethmoid region
* polyps in nasal cavity or the middle meatus, and/or
* radiographic imaging showing inflammation of the paranasal sinuses

Exclusion Criteria:

* Children
* Pregnant women (pregnancy test will be performed in women with child bearing potential)
* A mental condition rendering the subject unable to understand the nature, scope and possible consequences of the study
* Use of nasal or systemic corticosteroids or immunosuppressants 2 weeks prior to their visit
* Patients with cystic fibrosis or immunosuppression.
* Severe anatomic variations or deviations that do not allow access to all areas in the nasal cavity

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2021-07-25 (Actual); Study Completion 2021-07-25 (Actual)

PRIMARY OUTCOMES:
Nasal microbiome | 1 year
  Differences in microbial community composition between patients with N-ERD, CRSsNP, CRSwNP and healthy controls will be determined by 16S rRNA gene amplicon sequencing

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No